CLINICAL TRIAL: NCT04635332
Title: Effectiveness of a Combined Food Literacy and Physical Activity Intervention to Optimize Metabolic Health Among Women of Reproductive Age in Urban Uganda
Brief Title: Food Literacy and Physical Activity Intervention to Optimize Metabolic Health Among Women in Urban Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: VLIR-UOS (Unknown); Kyambogo University (Other); Our Lady of Africa Mbuya Catholic Parish (Unknown)
Responsible Party: Principal Investigator, Peter Yiga, PhD fellow, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS974ES
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Intervention Model Description: The intervention will be delivered through institutional religious women groups. A collaboration has been established with Our Lady of Africa Parish, Mbuya. Mbuya Catholic Parish has six sub parishes. These sub parishes will act as the clusters and will be the unit of randomization. The six sub parishes will be randomized to treatment and control arms. The six sub parishes (clusters) will be listed alphabetically. A cluster randomization with a 1:1 allocation will then be applied to randomize the sub parishes to either the treatment or control arm.
Who Masked: Participant
Masking Description: In the sub parishes, women group leaders and participants will be blinded about the study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the intervention arm, participants will be exposed to the developed intervention materials and face to face group sessions.
  Interventions: Behavioral: Food literacy and physical activity promotion interactive group sessions + Developed health promotion intervention materials (booklet)
- Control arm (Active Comparator): In the control arm, participants will only be given the developed intervention materials. Face to face group sessions will not be held for the control arm.
  Interventions: Behavioral: Developed health promotion intervention materials (booklet).

INTERVENTIONS:
Behavioral: Food literacy and physical activity promotion interactive group sessions + Developed health promotion intervention materials (booklet) — Information, skills training, goal setting and feedback interactive group sessions to improve food literacy aimed at increasing consumption of fruits and vegetables
  Information, skills training, goal setting and feedback interactive group sessions to increase engagement in moderate physical activity
  Information and skills training to increase ability to evaluate nutrition information
  In general, focus will be on increasing knowledge, skills and self-efficacy to develop a lifelong healthy and gastronomic relationship with food and physical activity.
  Arms: Intervention
Behavioral: Developed health promotion intervention materials (booklet). — In the control arm, participants will only be given the developed intervention materials (designed in form of the usual awareness programs). No group sessions will be conducted
  Arms: Control arm

SUMMARY:
Over the last 20 years, metabolic health (blood glucose and fats) of Ugandans, particularly residing in urban areas has increasingly become sub optimal. Women are the most affected. Sub optimal metabolic health increases chances of developing diseases known as non-communicable diseases (NCD); for example, type 2 diabetes and heart diseases. NCD are expensive to treat and Uganda lacks the health system to manage them. Therefore, there is need to prevent NCD. Metabolic health is mainly linked to dietary and physical activity behaviour. Studies show an increase in physical inactivity in urban Uganda, especially among women. Likewise, what urban Ugandans eat deviates from healthy recommendations by World Health Organization. For example, 9 in 10 urban Ugandans do not meet the daily fruit and vegetable health recommendations. Research shows that unhealthy eating and physical inactivity behaviours in urban Uganda are due to socio-cultural conceptions (prestige linked to weight gain and consumption of animal protein) and knowledge/skills gaps. Following the intervention mapping protocol, investigators have therefore designed an intervention to help women living in urban Uganda improve eating and physical activity behaviours to align them to healthy recommendations. Investigators target women because they are the most vulnerable health wise; possibility of passing on NCD risk from the mother to the offspring. Women are as well the most strategic for family behavioural change as they oversee dietary decisions in homes. The purpose of this study is to assess the effectiveness of a combined food literacy and physical activity intervention in optimizing metabolic health among women of reproductive age living in Urban Uganda. The study is a cluster randomized control trail divided into two phases: a three months intervention and a three months post-intervention follow-up phase. Primary outcome is waist circumference. The target group are women of reproductive age (18 to 45 years), residing in Kampala. Intervention will be delivered through religious women group structures.

DETAILED DESCRIPTION:
The study will be a cluster-randomized controlled trial. The CONSORT recommendations for cluster randomized trials will be followed (29). The study period is divided into two phases: a three months intervention and a three months post-intervention follow-up phase. The intervention will be delivered through institutional religious women groups. A collaboration has been established with Our Lady of Africa Parish, Mbuya. Mbuya Catholic Parish has six sub parishes. These sub parishes will act as the clusters and will be the unit of randomization. Within the sub parishes, there are existing women groups. These existing groups will be utilized for face to face intervention group sessions. For the intervention purposes, each group will be limited to a maximum of 14 members.

Intervention

In the intervention arm, participants will be exposed to the developed intervention materials (booklet) and face to face group sessions. In the group session, focus will be on increasing knowledge, skills and self-efficacy to develop a lifelong healthy and gastronomic relationship with food and physical activity. Specifically, the intervention will focus on increasing; women's ability to evaluate nutrition information; consumption of fruits and vegetables; and engagement in moderate physical activity. Investigators will provide information, skills training and feedback through monitoring. The intervention consists of five interactive group sessions. The group sessions will be two hours in length. In summary, the intervention will include;

* Profiling of personal gaps/needs; based on the baseline measurements, participants will be guided to compare their personal profiles (physical activity and fruit and vegetable intake) with WHO health recommendations,
* From this profiling, participants will brainstorm barriers and solutions to gaps in personal profile compared to health recommendations,
* Participants will then be guided to identify opportunities within their environment to improve personal profile, set personal SMART goals, and to come up with action plans to attain the set goals,
* Periodic feedback sessions aimed at reviewing and adapting the goals will be given. During feedback sessions, role models (participants who attain their goals) will share their experiences; challenges and enabling factors to motivate the other group members.

Vegetable recipes, practical tips to improve; food literacy, fruit and vegetable consumption and physical activity levels will be provided. The sessions will be moderated by a research team led by a PhD student who is trained in motivational interviewing.

Control arm

In the control arm, participants will only be given the developed intervention materials. Face to face group sessions will not be held for the control arm. Therefore, the research team will interface with the control groups at three moments; baseline measurements/distribution of developed intervention materials to the participants (designed in form of the usual awareness programs), post intervention measurements and post follow-up measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Sex (women)
2. Age (18 to 45 years)
3. Diagnosed with central obesity [waist circumference ≥ 80 cm]
4. Willingness to follow the three-months intervention and three months follow-up.
5. Willingness to participate in the study and to sign the informed consent

Exclusion Criteria:

1. Participants diagnosed or being treated for diabetes Mellitus Type 1 or Type 2
2. Participants being treated for hypertension, high cholesterol or any other cardio-metabolic related disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Waist circumference | Measured at baseline, at post intervention (at 3 months) and at post follow-up (at 6 months)
  Decreases in waist circumference are recommended as critically important treatment target for reducing adverse cardiometabolic health risks. Independent of sex and age, lifestyle induced reductions in waist circumference are associated with improvements in cardiometabolic risk factors with or without corresponding weight loss. Clinically relevant reductions in waist circumference can be achieved by routine, moderate- intensity exercise and/or dietary interventions consistent with WHO health recommendations. Thus, for the assessment of the effectiveness of lifestyle changes in adults, waist circumference is recommended. Waist circumference (to the nearest 0.5 cm) will be measured using a non-stretchable standard tape measure

SECONDARY OUTCOMES:
Fasting glucose, | Measured at baseline, at post intervention (at 3 months) and at post follow-up (at 6 months)
  CardioChek Plus will be used to assess the blood glucose
Lipid profile (total cholesterol, HDL cholesterol and triglycerides) | Measured at baseline, at post intervention (at 3 months) and at post follow-up (at 6 months)
  CardioChek Plus will be used to assess the lipid profile (total cholesterol, HDL, LDL and triglycerides).
Body composition | Measured at baseline, at post intervention (at 3 months) and at post follow-up (at 6 months)
  Body composition will be measured using Bodystat 1500 lite touch
Blood pressure | Measured at baseline, at post intervention (at 3 months) and at post follow-up (at 6 months)
  Blood pressure will be measured using blood pressure monitor - Seca b12
BMI | Height will be measured at baseline while weight will be measured at baseline, at post intervention (at 3 months) and at post follow-up (at 6 months)
  Height will be taken to the nearest 0.1 cm using a Seca digital height board. Weight will be measured to the nearest 0.1 kg using the Seca 874 dr.
Food literacy and fruit and vegetable intake | Measured at baseline, at post intervention (at 3 months) and at post follow-up (at 6 months)
  Food literacy will be assessed using the Ugandan food literacy questionnaire
Physical activity levels | Measured at baseline, at post intervention (at 3 months) and at post follow-up (at 6 months)
  Physical activity will be measured using the validated short form of the international physical activity questionnaire

OTHER OUTCOMES:
Process evaluation indicators (reach, dose and fidelity of intervention) | Assessed throughout the 3 months intervention
  Adherence to the programme

CONTACTS AND LOCATIONS:
Overall Officials: Peter Yiga, Principal Investigator — KU Leuven; Christophe Matthys, Study Chair — KU Leuven; Patrick Ogwok, Study Chair — Kyambogo University
Locations (1):
- Peter Yiga, Kampala, Uganda

REFERENCES:
- [Background] Yiga P, Seghers J, Ogwok P, Matthys C. Determinants of dietary and physical activity behaviours among women of reproductive age in urban sub-Saharan Africa: a systematic review. Br J Nutr. 2020 Oct 28;124(8):761-772. doi: 10.1017/S0007114520001828. Epub 2020 May 28. PMID 32460934
- [Background] Yiga P, Ogwok P, Achieng J, Auma MD, Seghers J, Matthys C. Determinants of dietary and physical activity behaviours among women of reproductive age in urban Uganda, a qualitative study. Public Health Nutr. 2021 Aug;24(12):3624-3636. doi: 10.1017/S1368980020003432. Epub 2020 Oct 1. PMID 33000718
- [Background] Ross R, Neeland IJ, Yamashita S, Shai I, Seidell J, Magni P, Santos RD, Arsenault B, Cuevas A, Hu FB, Griffin BA, Zambon A, Barter P, Fruchart JC, Eckel RH, Matsuzawa Y, Despres JP. Waist circumference as a vital sign in clinical practice: a Consensus Statement from the IAS and ICCR Working Group on Visceral Obesity. Nat Rev Endocrinol. 2020 Mar;16(3):177-189. doi: 10.1038/s41574-019-0310-7. Epub 2020 Feb 4. PMID 32020062
- [Background] Vidgen HA, Gallegos D. Defining food literacy and its components. Appetite. 2014 May;76:50-9. doi: 10.1016/j.appet.2014.01.010. Epub 2014 Jan 22. PMID 24462490
- [Background] Azevedo Perry E, Thomas H, Samra HR, Edmonstone S, Davidson L, Faulkner A, Petermann L, Manafo E, Kirkpatrick SI. Identifying attributes of food literacy: a scoping review. Public Health Nutr. 2017 Sep;20(13):2406-2415. doi: 10.1017/S1368980017001276. Epub 2017 Jun 27. PMID 28653598
- [Background] Eldredge LKB, Markham CM, Ruiter RA et al. (2016) Planning health promotion programs: an intervention mapping approach: John Wiley & Sons.
- [Derived] Yiga P, Van der Schueren B, Seghers J, Kiyimba T, Ogwok P, Tafiire H, Muluta SN, Matthys C. Effect of a complex lifestyle intervention to optimize metabolic health among females of reproductive age in urban Uganda, a randomized controlled trial. Am J Clin Nutr. 2023 Feb;117(2):436-443. doi: 10.1016/j.ajcnut.2022.12.005. Epub 2022 Dec 23. PMID 36811566
- [Derived] Yiga P, Van Lippevelde W, Seghers J, Ogwok P, Tafiire H, Muluuta SN, Matthys C. The conceptual framework for a combined food literacy and physical activity intervention to optimize metabolic health among women of reproductive age in urban Uganda. BMC Public Health. 2022 Feb 18;22(1):351. doi: 10.1186/s12889-022-12740-w. PMID 35183134